CLINICAL TRIAL: NCT01844115
Title: A Double-Blind, Placebo-Controlled, Flexible-Dose Study of Vilazodone in Patients With Generalized Anxiety Disorder.
Brief Title: Safety, Efficacy and Tolerability of Vilazodone in (GAD) Generalized Anxiety Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VLZ-MD-07
Record Dates: First submitted 2013-04-27; First posted 2013-05-01 (Estimated); Results first posted 2019-12-18 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-11

CONDITIONS: Generalized Anxiety Disorder
Keywords: Generalized Anxiety Disorder, GAD
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Vilazodone Hydrochloride; Administration, Oral

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Dose-matched placebo tablets, oral administration
  Interventions: Drug: Placebo
- Vilazodone (Experimental): Vilazodone tablets, oral administration
  Interventions: Drug: Vilazodone

INTERVENTIONS:
Drug: Placebo
  Other Names: Matching 10 mg and 20 mg placebo tablets, once-daily oral administration.
  Arms: Placebo
Drug: Vilazodone — Viibryd
  Other Names: Vilazodone, 20 mg once per day, oral administration, once daily or Vilazodone, 40 mg once daily, oral administration, once daily
  Arms: Vilazodone

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and tolerability of vilazodone relative to placebo in the treatment of generalized anxiety disorder (GAD).

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatient, 18-70 years of age
* Currently meet the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria for Generalized Anxiety Disorder
* Minimum score of 20 on Hamilton Rating Scale for Anxiety

Exclusion Criteria:

* Women who are pregnant or who will be breastfeeding during the study
* Patients with a history of:

  1. Any manic or hypomanic or mixed episode, including bipolar disorder and substance-induced manic, hypomanic or mixed episode
  2. Any depressive episode with psychotic or catatonic features
  3. Panic disorder with or without agoraphobia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 415 (Actual)
Dates: Start 2013-04-30 (Actual); Primary Completion 2014-03-31 (Actual); Study Completion 2014-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giovanna Forero, MA, Study Director — Forest Research Institute, a subsidiary of Actavis plc.
Locations (36):
- United States (36):
  - Forest Investigative Site 023, Birmingham, Alabama
  - Forest Investigative Site 013, Phoenix, Arizona
  - Forest Investigative Site 036, Beverly Hills, California
  - Forest Investigative Site 001, Costa Mesa, California
  - Forest Investigative Site 009, Oceanside, California
  - Forest Investigative Site 026, Rancho Mirage, California
  - Forest Investigative Site 017, Sherman Oaks, California
  - Forest Investigative Site 034, Sherman Oaks, California
  - Forest Investigative Site 030, Bradenton, Florida
  - Forest Investigative Site 029, Gainesville, Florida
  - Forest Investigative Site 035, Jacksonville, Florida
  - Forest Investigative Site 032, Orlando, Florida
  - Forest Investigative Site 021, West Palm Beach, Florida
  - Forest Investigative Site 025, Atlanta, Georgia
  - Forest Investigative Site 018, Decatur, Georgia
  - Forest Investigative Site 022, Hoffman Estates, Illinois
  - Forest Investigative Site 014, Berlin, New Jersey
  - Forest Investigative Site 005, Cherry Hill, New Jersey
  - Forest Investigative Site 015, Albuquerque, New Mexico
  - Forest Investigative Site 028, Brooklyn, New York
  - Forest Investigative Site 010, Brooklyn, New York
  - Forest Investigative Site 002, Cedarhurst, New York
  - Forest Investigative Site 004, Mount Kisco, New York
  - Forest Investigative Site 003, New York, New York
  - Forest Investigative Site 007, New York, New York
  - Forest Investigative Site 020, New York, New York
  - Forest Investigative Site 027, The Bronx, New York
  - Forest Investigative Site 019, Dayton, Ohio
  - Forest Investigative Site 008, Portland, Oregon
  - Forest Investigative Site 037, Allentown, Pennsylvania
  - Forest Investigative Site 011, Media, Pennsylvania
  - Forest Investigative Site 033, Memphis, Tennessee
  - Forest Investigative Site 031, Dallas, Texas
  - Forest Investigative Site 012, Herndon, Virginia
  - Forest Investigative Site 016, Bellevue, Washington
  - Forest Investigative Site 024, Seattle, Washington

REFERENCES:
- [Derived] Khan A, Durgam S, Tang X, Ruth A, Mathews M, Gommoll CP. Post Hoc Analyses of Anxiety Measures in Adult Patients With Generalized Anxiety Disorder Treated With Vilazodone. Prim Care Companion CNS Disord. 2016 Apr 28;18(2):10.4088/PCC.15m01904. doi: 10.4088/PCC.15m01904. eCollection 2016. PMID 27486544
- [Derived] Durgam S, Gommoll C, Forero G, Nunez R, Tang X, Mathews M, Sheehan DV. Efficacy and Safety of Vilazodone in Patients With Generalized Anxiety Disorder: A Randomized, Double-Blind, Placebo-Controlled, Flexible-Dose Trial. J Clin Psychiatry. 2016 Dec;77(12):1687-1694. doi: 10.4088/JCP.15m09885. PMID 27232052

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Vilazodone
Started | 202 | 202
Completed | 163 | 144
Not Completed | 39 | 58
Not completed — Adverse Event | 4 | 22
Not completed — Lack of Efficacy | 1 | 4
Not completed — Protocol Violation | 12 | 10
Not completed — Withdrawal by Subject | 11 | 11
Not completed — Lost to Follow-up | 11 | 10
Not completed — Pregnancy | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Population consisted of all patients in the Randomized Population who took at least 1 dose of double-blind investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Vilazodone | Total
Number analyzed (Participants) | 202 | 202 | 404
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.7 (13.4) | 39.2 (12.8) | 39.9 (13.1)
Age, Customized [Number; unit: Participants]
  < 20 | 4 | 2 | 6
  20-29 | 53 | 56 | 109
  30-39 | 42 | 55 | 97
  40-49 | 46 | 42 | 88
  50-59 | 36 | 26 | 62
  ≥ 60 | 21 | 21 | 42
Sex/Gender, Customized [Number; unit: Participants]
  Male | 65 | 75 | 140
  Female | 137 | 127 | 264
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 22 | 47
  Not Hispanic or Latino | 177 | 180 | 357
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 153 | 158 | 311
  Black or African American | 38 | 33 | 71
  Asian | 5 | 4 | 9
  American Indian or Alaska Native | 1 | 1 | 2
  Other | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Hamilton Rating Scale for Anxiety (HAM-A) Total Score
Description: The Hamilton Anxiety Rating Scale (HAM-A) is a clinician-administered scale which consists of 14 items, each rated on a five point scale ranging from 0 (not present) to 4 (very severe). The highest possible score is 56, which represents the most severe form of anxiety; the lowest possible score is 0, which represents an absence of anxiety.
Time Frame: Baseline to Week 8
Population: The Intent-to-Treat (ITT) Population consisted of all patients in the Safety Population who had at least 1 postbaseline assessment of the HAM-A.
Measure: Mean (Standard Deviation); unit: Score on Scale
Arm/Group | Placebo | Vilazodone
Number analyzed (Participants) | 200 | 200
Score on Scale | 14.7 (7.41) | 11.3 (6.99)
Statistical Analysis 1: Comparison: Placebo vs Vilazodone; Test type: Superiority; p = 0.0048, MMRM; Least Squares Mean Difference = -2.20, 95% CI 2-sided [-3.72 to -0.68]

2. Secondary Outcome: Change From Baseline in the Sheehan Disability Scale (SDS) Total Score
Description: The Sheehan Disability Scale (SDS) is a 3-item clinician-rated questionnaire used to evaluate impairments in the domains of work, social life/leisure, and family life/home responsibility. All items are rated on an 11-point continuum (0 = no impairment to 10 = most severe) with the total SDS score ranging from 0 (no impairment) to 30 (most severe).
Time Frame: Baseline to Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Placebo | Vilazodone
Number analyzed (Participants) | 200 | 200
Score on scale | 9.2 (6.96) | 7.4 (6.96)
Statistical Analysis 1: Comparison: Placebo vs Vilazodone; Test type: Superiority; p = 0.0236, MMRM; Least Squares Mean Difference = -1.89, 95% CI 2-sided [-3.52 to -0.26]

ADVERSE EVENTS:
Time Frame: Adverse events were collected until week 8.
Description: The Safety Population consisted of all patients in the Randomized Population who took at least 1 dose of double-blind investigational product.
Arm/Group | Placebo | Vilazodone
All-Cause Mortality (participants affected / at risk) | 0/202 | 0/202
Serious Adverse Events (participants affected / at risk) | 0/202 | 3/202
Other Adverse Events (participants affected / at risk) | 81/202 | 115/202
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=202) | Vilazodone (N=202)
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Urinary tract infection, (Infections and infestations) | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1
Stab wound (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo (N=202) | Vilazodone (N=202)
Nausea (Gastrointestinal disorders) | 26 | 60
Diarrhoea (Gastrointestinal disorders) | 12 | 56
Dry mouth (Gastrointestinal disorders) | 12 | 12
Upper respiratory tract infection (Infections and infestations) | 11 | 5
Dizziness (Nervous system disorders) | 8 | 22
Headache (Nervous system disorders) | 36 | 22
Somnolence (Nervous system disorders) | 6 | 12
Insomnia (Psychiatric disorders) | 8 | 15
Ejaculation delayed + (Reproductive system and breast disorders) | 1/65 | 4/75
Erectile dysfunction + (Reproductive system and breast disorders) | 1/65 | 4/75

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this study will be the property of Forest Research Institute, Inc. An integrated clinical and statistical report will be prepared at the completion of the study. Publication of the results by the investigator will be subject to mutual agreement between the investigator and Forest Research Institute, Inc.